CLINICAL TRIAL: NCT02661178
Title: A Phase 1, Blinded, Randomized, Placebo Controlled, Parallel-Group, Single-Dose, Dose-Escalation Study to Investigate Safety, Tolerability, and Pharmacokinetics of Emodepside (BAY 44-4400) After Oral Dosing in Healthy Male Subjects
Brief Title: First in Man Clinical Trial of Emodepside (BAY 44-4400)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Bayer (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DNDI-EMO-001; 2015-003592-29 (EudraCT Number)
Record Dates: First submitted 2016-01-15; First posted 2016-01-22 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: Parasitic Diseases; Helminthiasis; Nematode Infections; Secernentea Infections; Spirurida Infections; Filariasis; Skin Diseases, Parasitic; Skin and Connective Tissue Diseases; Skin Diseases; Skin Diseases, Infectious; Depsipeptides; Emodepside; Neglected disease; Africa; New drug; Oral drug; Parasite; Anthelmintic drug; Cyclooctadepsipeptide; Single ascending dose; Volunteers; Phase 1; Safety; Tolerability; Pharmacokinetics; Relative bioavailability; Onchocerciasis
MeSH Terms: conditions — Parasitic Diseases; Helminthiasis; Nematode Infections; Secernentea Infections; Spirurida Infections; Filariasis; Skin Diseases, Parasitic; Skin and Connective Tissue Diseases; Skin Diseases; Skin Diseases, Infectious; Neglected Diseases; Onchocerciasis | interventions — emodepside; Bay 44-4400

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- emodepside (BAY 44-4400) (Experimental): Up to 10 cohorts with single ascending dose
  Interventions: Drug: emodepside (BAY 44-4400)
- placebo of emodepside (BAY 44-4400) (Placebo Comparator): Up to 10 cohorts with single ascending dose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: emodepside (BAY 44-4400)
  Arms: emodepside (BAY 44-4400)
Drug: placebo
  Arms: placebo of emodepside (BAY 44-4400)

SUMMARY:
This study will investigate the safety, tolerability, and pharmacokinetics of single ascending doses of emodepside (BAY 44-4400) in healthy male volunteers. This study will also conduct an exploratory investigation of the relative bioavailability of emodepside administered as tablets and determine the effect of food on the pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Male, Caucasian volunteers, deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine. Optionally, after further evaluation during the study, at the sponsor's discretion other ethnic groups may be recruited.
* Aged 18 to 55 years.
* With a body mass index (BMI; Quetelet index) in the range of 18 to 30.1 kg/m2 at screening.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate, after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate

Exclusion Criteria:

* Participation in another clinical trial within 3 months prior and during the study, or 5-times the half-life of the drug tested in the previous clinical trial, whichever is longer (time calculated relative to the last dose in the previous clinical trial)
* Clinically relevant abnormal medical history, concurrent medical condition, acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of study drug taken orally.
* Presence of abnormal physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the subject.
* Positive tests for hepatitis B & C, HIV
* Presence or history of drug or alcohol abuse during the last 10 years, or intake of more than 21 units of alcohol weekly.
* Regular daily consumption of more than one liter of xanthine-containing beverages
* Regular daily consumption of more than 5 cigarettes daily, or use more than 3 grams (1/8 ounce) of tobacco
* Use of a prescription medicine during the 28 days before the first dose of trial medication or use of an over-the-counter medicine, with the exception of acetaminophen (paracetamol), during the 7 days before the first dose of trial medication
* Use of dietary supplements or herbal remedies (such as St John's Wort) known to interfere with the CYP3A4 and/or P-gp metabolic pathways during the 28 days before the first dose of trial medication (see list in Study Procedures Manual)

Additional exclusion criteria for cohort with ophthalmological assessments:

* No contact lenses wear within 1 month prior to first dose of IMP. Contact lenses wear is not permitted during the study
* Any ocular disorder for which topical ocular therapy is currently or chronically prescribed, including inflammatory eye disease (dry eye allergic conjunctivitis [seasonal allergic conjunctivitis, vernal keratoconjunctivitis, atopic keratoconjunctivitis], uveitis and glaucoma)
* Past history of ocular disease requiring ongoing treatment
* Past ocular surgery including laser or other refractive corneal surgery
* Evidence of eye irritation, visual difficulties, corneal opacity, ocular surface (corneal or conjunctival damage, with or without ocular symptoms)
* Evidence of narrow anterior chamber angles causing increased risk of acute glaucoma
* Evidence of ocular media opacity including lens opacity/vitreous opacities
* Evidence of retinal or optic nerve pathology
* Evidence of pronounced colour blindness, as indicated by an Ishihara score of 9/13 or below

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, MD, BSc, Principal Investigator — Hammersmith Medicines Research; Frederic Monnot, Study Director — Drugs for Neglected Diseases initiative
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 79 healthy subjects were randomized and received study drug. Protocol Enrollment reflects the total number of participants enrolled in both Part 1 (63 participants) and Part 2 (16 participants).
Groups:
- Emodepside 0.1mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 0.1mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 1mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 1mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 2.5mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 2.5mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 5mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 5mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 5mg Tablet, Fasted (Part 1): Emodepside (BAY 44-4400) 5mg tablet (immediate release), administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 10mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 10mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 20mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 20mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 20mg Tablet, Fasted (Part 1): Emodepside (BAY 44-4400) 20mg tablet (immediate release), administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 40mg Solution, Fasted (Part 1): Emodepside (BAY 44-4400) 40mg solution, as oral liquid service formulation, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Placebo Solution, Fasted (Part 1): Matching placebo of emodepside (BAY 44-4400), solution, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Placebo Tablet, Fasted (Part 1): Matching placebo of emodepside (BAY 44-4400), tablet, administered in fasted state Part one of study (FIH, single ascending dose phase)
- Emodepside 10mg Solution, Fed (Part 2): Emodepside (BAY 44-4400) 10mg solution, as oral liquid service formulation, administered in fed state This cohort was not classed as first in human Part two of study (not FIH, exploratory effect of food on the bioavailability of emodepside and to assess relationship between emodepside and adverse events)
- Emodepside 40mg Solution, Fasted, (Part 2): Emodepside (BAY 44-4400) 40mg solution, as oral liquid service formulation, administered in fasted state Part two of study (not FIH, exploratory effect of food on the bioavailability of emodepside and to assess relationship between emodepside and adverse events)
- Placebo Solution, Fed (Part 2): Matching placebo of emodepside (BAY 44-4400), solution, administered in fed state Part two of study (not FIH, exploratory effect of food on the bioavailability of emodepside and to assess relationship between emodepside and adverse events)
- Placebo Solution, Fasted (Part 2): Matching placebo of emodepside (BAY 44-4400), solution, administered in fasted state Part two of study (not FIH, exploratory effect of food on the bioavailability of emodepside and to assess relationship between emodepside and adverse events)
Period: Part 1
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Started | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Emodepside 40mg Solution, Fasted, AE Follow-up Arm (Part 2): Emodepside (BAY 44-4400) 40mg solution, as oral liquid service formulation, administered in fasted state Part two of study (not FIH, exploratory effect of food on the bioavailability of emodepside and to assess relationship between emodepside and adverse events)
- Total: Total of all reporting groups
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, AE Follow-up Arm (Part 2) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2) | Total
Number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 6 | 6 | 2 | 2 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Totals were calculated seperately for Parts 1 and 2
  years
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1 | 23 (0) | 38.6 (10.06) | 34.8 (9.20) | 29.3 (8.12) | 36.8 (10.69) | 34.2 (10.55) | 32.8 (9.75) | 31.3 (8.91) | 30.8 (10.83) | 30.7 (7.46) | 28.0 (3.56) |  |  |  |  | 32.4 (8.89)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2 |  |  |  |  |  |  |  |  |  |  |  | 27.7 (7.34) | 38.5 (10.67) | 51.5 (0.71) | 40 (11.31) | 38.3 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Totals were calculated seperately for Parts 1 and 2
  Participants
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 1: Male | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 |  |  |  |  | 63
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2: Female |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part 2: Male |  |  |  |  |  |  |  |  |  |  |  | 6 | 6 | 2 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Totals were calculated seperately for Parts 1 and 2
  Participants
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 |  |  |  |  | 3
    Part 1: Not Hispanic or Latino | 1 | 5 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 11 | 3 |  |  |  |  | 60
    Part 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2: Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  | 1 | 0 | 0 | 0 | 1
    Part 2: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  | 5 | 6 | 2 | 2 | 15
    Part 2: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Totals were calculated seperately for Parts 1 and 2
  Participants
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 1: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 1: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 1: White | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 |  |  |  |  | 63
    Part 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part 2: Asian |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part 2: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part 2: Black or African American |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part 2: White |  |  |  |  |  |  |  |  |  |  |  | 6 | 6 | 2 | 2 | 16
    Part 2: More than one race |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part 2: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Population: Totals were calculated seperately for Parts 1 and 2
  cm
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1 | 173 (0) | 176.8 (4.87) | 179.8 (6.24) | 175.5 (5.82) | 177.2 (10.87) | 177.2 (3.54) | 179.0 (7.51) | 179.5 (7.45) | 183.3 (7.63) | 180.0 (7.98) | 183.3 (2.99) |  |  |  |  | 179.1 (6.89)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2 |  |  |  |  |  |  |  |  |  |  |  | 183.2 (6.37) | 176.0 (5.22) | 178 (8.49) | 181 (4.24) | 179.6 (6.28)
Weight [Mean (Standard Deviation); unit: kg] — Population: Totals were calculated seperately for Parts 1 and 2
  kg
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1 | 72.00 (0) | 70.64 (6.815) | 75.47 (11.331) | 75.83 (3.506) | 76.56 (13.197) | 74.80 (11.383) | 81.93 (10.397) | 81.73 (9.075) | 83.27 (11.267) | 79.52 (10.130) | 85.15 (7.217) |  |  |  |  | 78.43 (9.931)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2 |  |  |  |  |  |  |  |  |  |  |  | 82.20 (7.979) | 82.65 (13.598) | 72.8 (1.98) | 83.7 (24.75) | 81.38 (11.636)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Totals were calculated seperately for Parts 1 and 2
  kg/m^2
    Part 1: number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 4 | 0 | 0 | 0 | 0 | 63
    Part 1 | 24.10 (0) | 22.60 (2.117) | 23.30 (2.683) | 24.65 (1.162) | 24.20 (1.707) | 23.75 (2.868) | 25.55 (2.651) | 25.43 (3.169) | 24.72 (2.613) | 24.49 (2.131) | 25.38 (2.291) |  |  |  |  | 24.41 (2.356)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 2 | 2 | 16
    Part 2 |  |  |  |  |  |  |  |  |  |  |  | 24.5 (2.137) | 26.55 (3.213) | 23.1 (2.83) | 25.4 (6.36) | 25.21 (3.117)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Measured by Adverse Events
Description: Deaths, serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs)
Time Frame: Up to 14 days post dose (may be extended to 21 days)
Population: AEs were determined in the Safety Population. In Part 1 n=63 (n=62 subjects completed). One subject in the 1mg emodepside group was withdrawn after receiving 0.1mg emodepside LSF, owing to an AE. He consented to follow-up safety assessment until Day 7 as a 0.1mg emodepside group.
  In Part 2, n=16 (n=16 subjects completed)
Measure: Number; unit: participants
Groups:
- Emodepside 0.1mg Solution, Fasted (Part 1): No AEs were reported for Emodepside (BAY 44-4400) 0.1mg solution, as oral liquid service formulation, administered in fasted state
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 2 | 2
participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subjects with SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subjects with TEAE | 1 | 3 | 0 | 3 | 3 | 5 | 3 | 2 | 5 | 3 | 5 | 5 | 1 | 0 | 0

2. Primary Outcome: Safety and Tolerability as Measured by Physical and Neurological Examination Findings
Description: Abnormal or clinically significant neurological examination findings during the study or reported as an AE
Time Frame: Up to 14 days post dose (may be extended to 21 days)
Population: AEs were determined in the Safety Population. In Part 1 n=63 (n=62 subjects completed). One subject in the 1mg emodepside group was withdrawn after receiving 0.1mg emodepside LSF, owing to an AE. He consented to follow-up safety assessment until Day 7 as a 0.1mg emodepside group.
Measure: Number; unit: participants
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 2 | 2
participants
  Abnormal neurological examination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neurological examination reported as AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal physcial examination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Physical examination reported as AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Safety and Tolerability as Measured by Vital Signs
Description: Vital signs included heart rate, systolic and diastolic blood pressure,
Time Frame: Up to 14 days post dose (may be extended to 21 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 2 | 2
participants
  Clinically significant change in heart rate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically significant change in systolic BP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically significant change in diastolic BP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Safety and Tolerability as Measured by 12-lead ECG
Description: The following variables were recorded in 12-lead ECGs and extracted from continuous 12-lead ECG recordings: ventricular rate, PR interval, QRS interval, QTcB and QTcF interval.
Time Frame: Up to 14 days post dose (may be extended to 21 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 2 | 2
participants
  Notable changes in ventricular rate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Notable changes in PR interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Notable changes in QRS interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Notable changes in QTcB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Notable changes in QTcF interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Safety and Tolerability as Measured by Clinical Laboratory Parameters
Description: Clinical laboratory parameters included hematology, biochemistry, serology and coagulation in blood samples and urinalysis in urine samples
Time Frame: Up to 14 days post dose (may be extended to 21 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
Number analyzed (Participants) | 1 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 2 | 2
participants
  Clinically significant hematological changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically significant biochemical changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically significant serological changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically significant coagulation changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically significant urinalysis changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Safety and Tolerability as Measured by Ophthalmological Examination Findings in One Study Arm Only
Description: Subjects attended a specialist eye hospital for ophthalmology assessments by a Consultant Ophthalmologist. Opthalmology assessments included:ocular symptoms, past ocular history, auto-refraction, best corrected distance visual acuity, color vision assessment, amsler grid assessment, ocular alignment and ocular motility assessment, confrontation visual field assessment, slit lamp examination (anterior segment), intraocular pressure (Goldmann Tonometry), optical coherence scanning of tomography, post mydriatic ocular media (at Screening visit 2 only) and retinal examination with slit lamp and lens.
Time Frame: Up to 14 days post dose (may be extended to 21 days)
Population: AEs were determined in the Safety Population. Opthalmology examinations were only performed for the Emodepside 40mg group (n=6) and the corresponding placebo group (n=2)
Measure: Number; unit: participants
Arm/Group | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 2)
Number analyzed (Participants) | 6 | 2
participants
  Clinically significant occular symptoms | 4 | 0
  Clinically significant best corrected vis acuity | 1 | 0
  Clinically significant changes in remaining exams | 0 | 0

7. Secondary Outcome: The AUC∞ of Emodepside in Plasma
Description: The area under the plasma drug concentration versus time curve from time zero to infinity (AUC∞)
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: It is unacceptable to use AUCinf data if>40% of the AUC has been extrapolated.This is in line with literature(Gabrielson&Weiner, 2000).The AUCinf values with<20% of the area extrapolated (reliable results) have not been summarised in the tables because n is either 1 or 2 per treatment (n=2 only for 1m solution).
Measure: Geometric Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 1
h*ng/ml | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above | NA (NA) — see explanation above

8. Secondary Outcome: The AUC∞/D of Emodepside in Plasma
Description: Dose-normalized area under the plasma drug concentration versus time curve from time zero to infinity (AUC∞/D), calculated as AUC∞/Dose administered.
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 7
Measure: Number; unit: No values calculated
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 1
No values calculated | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above | NA — see explanation above

9. Secondary Outcome: The Cmax of Emodepside in Plasma
Description: Maximum observed plasma concentration (Cmax) was obtained directly from the concentration-time data
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: PK Concentration were summarized using PK concentration population (all subjects who received at least one dose of study drug and for whom a PK sample was analyzed). PK parameters were summarized using the PK Parameter population (all subjects in the PK Concentration Population for whom PK parameters could be derived).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
ng/mL | 18.6 (20.8) | 37.6 (15.5) | 92.1 (16.2) | 25.7 (23.9) | 172 (32.3) | 306 (28.7) | 30.2 (62.5) | 595 (27.9) | 71.9 (29.6) | 434 (32.7) |

10. Secondary Outcome: The Cmax/D of Emodepside in Plasma
Description: Dose-normalized observed maximum plasma concentration (Cmax/D) was calculated as Cmax/Dose administered
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: PK Concentration data were summarized using the PK concentration population (all subjects who received at least one dose of study drug and for whom a PK sample was analyzed). PK parameters were summarized using the PK Parameter population (all subjects in the PK Concentration Population for whom PK parameters could be derived).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
(ng/mL)/mg | 18.6 (20.8) | 15.0 (15.5) | 18.4 (16.2) | 5.15 (23.9) | 17.2 (32.3) | 15.3 (28.7) | 1.51 (62.5) | 14.9 (27.9) | 71.9 (29.6) | 10.9 (32.7) |

11. Secondary Outcome: The Cmax, Norm of Emodepside in Plasma
Description: The observed maximum plasma concentration (Cmax) normalized by dose and body weight was calculated as Cmax/(Dose administered*body weight)
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/(mg*kg)
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
(ng/mL)/(mg*kg) | 0.265 (25.1) | 0.203 (25.2) | 0.244 (18.4) | 0.0680 (27.7) | 0.233 (46.7) | 0.189 (35.7) | 0.0187 (69.1) | 0.178 (36.3) | 0.0882 (28.9) | 0.133 (49.7) |

12. Secondary Outcome: The Tmax of Emodepside in Plasma
Description: Time to reach maximum plasma concentration (Tmax) was obtained directly from the concentration-time data
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Mean (Full Range); unit: Hours
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
Hours | 1.00 [1.00 to 1.05] | 1.00 [1.00 to 2.50] | 1.00 [1.00 to 1.50] | 2.00 [1.02 to 2.55] | 1.00 [1.00 to 1.00] | 1.50 [1.00 to 2.53] | 2.00 [1.50 to 2.02] | 1.05 [1.00 to 8.00] | 2.50 [2.00 to 2.52] | 0.967 [0.950 to 3.00] |

13. Secondary Outcome: The t½ of Emodepside in Plasma
Description: Terminal half-life (t½), calculated according to the equation t½ = ln2/λz, where λz is the apparent terminal elimination rate constant, estimated by linear regression of log-transformed concentration versus time data
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
Hours | 42.7 (531) | 449 (74.0) | 415 (117) | 267 (392) | 365 (286) | 590 (68.1) | 348 (171) | 392 (31.7) | 531 (99.3) | 440 (49.9) |

14. Secondary Outcome: The MRT of Emodepside in Plasma
Description: The mean residence time (MRT) was calculated as MRT = AUMC/AUC∞, where AUMC is the area under the first moment of the concentration-time curve from zero time (pre-dose) extrapolated to infinite time
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
Hours | 52.7 (528) | 572 (78.8) | 570 (92.1) | 337 (430) | 533 (232) | 757 (69.9) | 443 (182) | 489 (31.4) | 752 (91.7) | 569 (52.5) |

15. Secondary Outcome: The CL/F of Emodepside in Plasma
Description: Apparent total clearance from plasma (CL/F) was calculated as CL/F = Dose/AUC∞
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
L/hour | 3.88 (151) | 1.37 (44.1) | 1.34 (57.8) | 4.79 (179) | 1.42 (115) | 1.34 (24.8) | 13.3 (150) | 1.57 (32.6) | 1.42 (57.3) | 1.69 (22.1) |

16. Secondary Outcome: The AUC 0-24 of Emodepside in Plasma
Description: Area under the plasma concentration-time curve from time zero (pre-dose) to 24 h was calculated using the trapezoidal method
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
h*ng/mL | 100 (50.4) | 250 (6.50) | 522 (25.8) | 183 (24.3) | 996 (21.2) | 1910 (16.3) | 223 (58.0) | 4110 (33.6) | 673 (26.4) | 3320 (26.0) |

17. Secondary Outcome: The AUC 0-24/D of Emodepside in Plasma
Description: Dose-normalized area under the concentration-time curve (AUC) from time zero (pre-dose) to 24 h was calculated as AUC0-24/Dose administered
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h.ng/mL)/mg)
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
(h.ng/mL)/mg) | 100 (50.4) | 100 (6.50) | 104 (25.8) | 36.5 (24.3) | 99.6 (21.2) | 95.3 (16.3) | 11.2 (58.0) | 103 (33.6) | 67.3 (26.4) | 82.9 (26.0) |

18. Secondary Outcome: The AUC 24, Norm of Emodepside in Plasma
Description: Area under the concentration-time curve from time zero (pre-dose) to 24 h, normalized by dose and body weight (AUC 24, norm) was calculated as AUC0-24/(Dose administered*body weight)
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/(mg*kg)
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
(h*ng/mL)/(mg*kg) | 1.43 (58.7) | 1.35 (17.5) | 1.38 (27.8) | 0.483 (28.9) | 1.35 (33.8) | 1.18 (27.8) | 0.138 (66.0) | 1.23 (42.9) | 0.825 (30.8) | 1.01 (45.8) |

19. Secondary Outcome: The Vz/F of Emodepside in Plasma
Description: Apparent volume of distribution (Vz/F) was calculated as Vz/F = Dose/(λz × AUC∞), where λz is the apparent terminal elimination rate constant, estimated by linear regression of log-transformed concentration versus time data
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
Litres | 239 (88.0) | 885 (27.4) | 802 (49.1) | 1850 (56.1) | 748 (68.7) | 1140 (47.1) | 6700 (40.1) | 888 (21.3) | 1090 (36.2) | 1070 (41.8) |

20. Secondary Outcome: The AUC Last of Emodepside in Plasma
Description: The area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration (t), calculated using the linear trapezoidal method for increasing concentrations and the log trapezoidal method for decreasing concentrations
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
h*ng/mL | 182 (111) | 845 (10.4) | 1700 (24.2) | 501 (76.8) | 3070 (27.7) | 7480 (22.1) | 667 (125) | 16400 (23.6) | 3390 (20.4) | 13800 (23.4) |

21. Secondary Outcome: Frel of the IR (Immediate Release) Tablet of Emodepside
Description: The average relative bioavailability (Frel) of the IR tablet was calculated
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: Frel percentage
Groups:
- Emodepside 5mg Solution Versus Tablet, Fasted (Part 1): Emodepside (BAY 44-4400) 5mg solution versus tablet, administered in fasted state Part one of study
- Emodepside 20mg Solution Versus Tablet, Fasted (Part 1): Emodepside (BAY 44-4400) 20mg solution versus tablet, administered in fasted state Part one of study
Arm/Group | Emodepside 5mg Solution Versus Tablet, Fasted (Part 1) | Emodepside 20mg Solution Versus Tablet, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6
Frel percentage | 35.0 [26.6 to 46.0] | 11.7 [7.73 to 17.8]

22. Secondary Outcome: The AUC Last, Norm of Emodepside in Plasma
Description: The area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration normalized by dose and body weight (AUClast/(Dose administered*body weight))
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/(mg*kg)
Arm/Group | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Emodepside 0.1mg Solution, Fasted (Part 1)
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 0
(h*ng/mL)/(mg*kg) | 2.60 (127) | 4.56 (19.5) | 4.50 (27.1) | 1.33 (78.4) | 4.17 (42.6) | 4.62 (30.8) | 0.414 (138) | 4.91 (36.5) | 4.16 (25.5) | 4.21 (42.6) |

23. Secondary Outcome: Effect of Food on the Bioavailability (Cmax) of Emodepside (BAY 44-4400) After Single Oral Dose Administered as Solution or IR Tablets in One Arm Only
Description: Results of the statistical analysis of the effect of food on Emodepside exposure, after a single dose of 10 mg Emodepside LSF solution.
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: emodepside assessed in fasted condition: only one cohort (10mg solution) assessed with high fat high calories meal.
Measure: Least Squares Mean (Full Range); unit: ng/ml
Groups:
- Emodepside 10mg Solution Fasted: Emodepside (BAY 44-4400) 10mg solution, as oral liquid service formulation, administered in fasted state
- Emodepside 10mg Solution Fed: Emodepside (BAY 44-4400) 10mg solution, as oral liquid service formulation, administered in fed state
Arm/Group | Emodepside 10mg Solution Fasted | Emodepside 10mg Solution Fed
Number analyzed (Participants) | 6 | 6
ng/ml | 172 [96.7 to 227.0] | 71.9 [47.4 to 109.0]

24. Secondary Outcome: Effect of Food on the Bioavailability (AUC24) of Emodepside (BAY 44-4400) After Single Oral Dose Administered as Solution or IR Tablets in One Arm Only
Description: as for outcome 23
Time Frame: From pre-dose until 336h post-dose (may be extended to 504h post-dose)
Population: emodepside assessed in fasted condition: only one cohort (10mg solution) assessed with high fat high calories meal.
Measure: Least Squares Mean (Full Range); unit: ng*h/mL
Arm/Group | Emodepside 10mg Solution Fasted | Emodepside 10mg Solution Fed
Number analyzed (Participants) | 6 | 6
ng*h/mL | 996 [753 to 1380] | 673 [520 to 982]

ADVERSE EVENTS:
Time Frame: The AE reporting period for this trial began after subject enrolment in the trial (after signature of informed consent) and ended at the follow-up visit (3 weeks after their dose of study medicine) .
Arm/Group | Emodepside 0.1mg Solution, Fasted (Part 1) | Emodepside 1mg Solution, Fasted (Part 1) | Emodepside 2.5mg Solution, Fasted (Part 1) | Emodepside 5mg Solution, Fasted (Part 1) | Emodepside 5mg Tablet, Fasted (Part 1) | Emodepside 10mg Solution, Fasted (Part 1) | Emodepside 20mg Solution, Fasted (Part 1) | Emodepside 20mg Tablet, Fasted (Part 1) | Emodepside 40mg Solution, Fasted (Part 1) | Emodepside 10mg Solution, Fed (Part 2) | Emodepside 40mg Solution, Fasted, (Part 2) | Placebo Solution, Fasted (Part 1) | Placebo Tablet, Fasted (Part 1) | Placebo Solution, Fed (Part 2) | Placebo Solution, Fasted (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/4 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/4 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 3/5 | 0/6 | 3/6 | 3/5 | 5/6 | 3/6 | 2/6 | 5/6 | 3/6 | 5/6 | 5/12 | 1/4 | 0/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Emodepside 0.1mg Solution, Fasted (Part 1) (N=1) | Emodepside 1mg Solution, Fasted (Part 1) (N=5) | Emodepside 2.5mg Solution, Fasted (Part 1) (N=6) | Emodepside 5mg Solution, Fasted (Part 1) (N=6) | Emodepside 5mg Tablet, Fasted (Part 1) (N=5) | Emodepside 10mg Solution, Fasted (Part 1) (N=6) | Emodepside 20mg Solution, Fasted (Part 1) (N=6) | Emodepside 20mg Tablet, Fasted (Part 1) (N=6) | Emodepside 40mg Solution, Fasted (Part 1) (N=6) | Emodepside 10mg Solution, Fed (Part 2) (N=6) | Emodepside 40mg Solution, Fasted, (Part 2) (N=6) | Placebo Solution, Fasted (Part 1) (N=12) | Placebo Tablet, Fasted (Part 1) (N=4) | Placebo Solution, Fed (Part 2) (N=2) | Placebo Solution, Fasted (Part 2) (N=2)
TEAEs by primary system organ classes (SOCs) (Nervous system disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 4 | 2 | 0 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 5 | 0 | 5 | 0 | 1 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0
TEAEs by primary system organ classes (SOCs) (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TEAEs by primary system organ classes (SOCs) (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution (HMR) could not make any public communication related to the Results or Trial Subjects, notably, without DNDi's prior written approval. The Institution shall inform DNDi in advance of any media visits to the Clinical Trial site and comply with the guidance provided by DNDi.

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT02661178/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02661178/SAP_001.pdf